CLINICAL TRIAL: NCT00220493
Title: Clinical Study Protocol: Evaluation of the Efficiency of Ritalin in Multiple Sclerosis Patients
Brief Title: Evaluation of Efficiency of Ritalin in Multiple Sclerosis (MS) Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: SHEBA-03-2966-AA-CTIL
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive
Keywords: MS; RITALIN; PASAT; COGNITION; ATTENTION; Relapsing remitting; Secondary progressive; Primary progressive
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Methylphenidate

INTERVENTIONS:
Drug: Ritalin

SUMMARY:
Scientific background:

Growing awareness and accumulating data regarding the cognitive impairment and its progression in multiple sclerosis (MS) patients has received an important place in neurological research in the last decade.

DETAILED DESCRIPTION:
Scientific background:

Growing awareness and accumulating data regarding the cognitive impairment and its progression in multiple sclerosis (MS) patients has received an important place in neurological research in the last decade. Cognitive impairments occur frequently (43 to 65%) in MS. Moreover, in up to 50% of patients in whom no cognitive disturbances are found on routine neurological examination, cognitive impairments can be elicited using sensitive and disease specific neuropsychological tests. Even in patients with short disease duration of less than two years, discrete impairment of cognitive function may be found in up to 60% on neuropsychological testing without impacting activities of daily living.

We have recently reported that cognitive impairment occurred in 53.7% of patients with probable MS (evaluated within a mean of one month of the onset of new neurological symptoms). Verbal abilities and attention span were most frequently affected (43.3 and 41.8% respectively). An additional study demonstrated that MS patients within the first 5 years of disease onset presented attentional dysfunction only when the cognitive load of the attention task was high and when controlled information processing was required. This high rate of attention impairment found in MS patients early in the disease process may have a significant impact on quality of life and activities of daily living as attention is one of the most fundamental cognitive functions essential for normal daily activities and a requisite step towards conscious perception. Consequently, we suggest investigating whether treatment with Ritalin (methylphenidate) has an effect on patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite MS according to Poser criteria;
* Attention impairment defined as abnormal PASAT score;
* Written and signed informed consent;

Exclusion Criteria:

* Pregnancy or lactation;
* Steroid treatment;
* Persistent psychostimulant treatment;
* MS relapse;

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-06; Study Completion 2005-06

PRIMARY OUTCOMES:
Score on the Paced Auditory Serial Addition Test (PASAT) one hour after taking the drug/placebo

CONTACTS AND LOCATIONS:
Overall Officials: Anat Achiron, MD PhD, Principal Investigator — Sackler School of Medicine; Yirmiyahu Harel, MD, Principal Investigator — Sachler School of Medicine; Nava Appleboim-Gavish, MA, Principal Investigator — Sheba Medical Center at Tel Hashomer Israel
Locations (1):
- Multiple Sclerosis Center, Ramat Gan, Israel